CLINICAL TRIAL: NCT02990325
Title: An Open-Label Study of the Safety, Pharmacokinetics, and Pharmacodynamics of ABX464 in HIV-1 Seronegative and Seropositive Adults
Brief Title: A Safety, Pharmacokinetics, and Pharmacodynamics Study of ABX464 in HIV-1 Seronegative and Seropositive Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Abivax S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABX464-005
Record Dates: First submitted 2016-12-07; First posted 2016-12-13 (Estimated); Results first posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: HIV Infections; Health Volunteers
Keywords: ABX464, HIV infection
MeSH Terms: conditions — HIV Infections | interventions — ABX464

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ABX464 150mg (Experimental): ABX464, 50mg per Capsule Three Capsules per day for 28 days
  Interventions: Drug: ABX464 150mg
- ABX464 50mg for 28 days (Experimental): ABX464, 50mg per Capsule One Capsule per day for 28 days
  Interventions: Drug: ABX464 50mg
- ABX464 50mg for 84 days (Experimental): ABX464, 50mg per Capsule One Capsule per day for 84 days
  Interventions: Drug: ABX464 50mg

INTERVENTIONS:
Drug: ABX464 150mg — ABX464 given orally at 150 mg per day from Day 0 to Day 28 (Cohort 1/ HIV infected subjects)
  Arms: ABX464 150mg
Drug: ABX464 50mg — ABX464 given orally at 50 mg per day from Day 0 to Day 28 (Cohort 2 / non HIV infected subjects)
  Arms: ABX464 50mg for 28 days
Drug: ABX464 50mg — ABX464 given orally at 50 mg per day from Day 0 to Day 84 (Cohort 3 / HIV infected subjects)
  Arms: ABX464 50mg for 84 days

SUMMARY:
The purpose of the ABX464-005 study is to characterize the systemic and mucosal immunological sequelae associated with exposure to ABX464 and to explore selected immunological endpoints, compartmental pharmacokinetics, and pharmacodynamics.

DETAILED DESCRIPTION:
The purpose of the ABX464-005 study is to characterize the systemic and mucosal immunological sequelae associated with exposure to ABX464 and to explore selected immunological endpoints, compartmental pharmacokinetics, and pharmacodynamics. The site will screen and enroll 12 HIV-infected subjects who will receive 150 mg ABX464 orally once daily for 28 days (Cohort 1). Following completion of this cohort a further 24 subjects will be enrolled: 12 HIV-uninfected subjects will receive 50 mg ABX464 orally once daily for 28 days (Cohort 2) and 12 HIV-infected subjects (Cohort 3) who will 50 mg ABX464 orally once daily for 84 days.

ELIGIBILITY:
Inclusion criteria:

* Males aged 18-65 years;
* Subjects with adequate hematological and biochemical laboratory parameters
* Subjects should be able and willing to comply with study visits and procedures as per protocol;
* Subjects should understand, sign and date the written voluntary informed consent form at the screening visit prior to any protocol-specific procedures being performed;
* Subjects must agree to use in addition to the condom, a second highly effective method (one for the subject and one for the partner) of contraception (defined as per the Clinical Trials Facilitation and Coordination Group (CTFG) Guidance).

For HIV positive Subjects

* Subjects with a positive HIV-1 serology at any time before the study entry.
* Subjects treated for at least 12 months prior to screening with Dolutegravir or Raltegravir combined with either Tenofovir + Emtricitabine (TDF/FTC) or Abacavir + Lamivudine (ABC/3TC);
* Subjects with HIV plasma viral load ≤ 50 copies/mL during the 6 months prior to screening with a maximum of 2 blips ≤ 1000 copies during this period;
* Subjects' HIV-1 plasma viral load to be ≤ 100,000 copies/mL at any time beyond 6 months after the estimated date of primary infection;

Exclusion Criteria:

* History of allergic disease, anaphylaxis or reactions likely to be triggered or exacerbated by any component of investigational products;
* Acute or chronic infectious disease other than HIV infection (include but not limited to viral hepatitis such as hepatitis B, hepatitis C, active tuberculosis, active syphilis [i.e. currently treated].
* Acute, chronic or history of clinically relevant pulmonary, cardiovascular, gastrointestinal, hepatic, pancreatic or renal functional abnormality, encephalopathy, neuropathy or unstable Central Nervous System (CNS) pathology, angina or cardiac arrhythmias, or any other clinically significant medical problems as determined by physical examination and/or laboratory screening tests and/or medical history;
* Severe hepatic impairment;
* Acute, chronic or history of immunodeficiency or autoimmune disease other than HIV infection;

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2018-12-27 (Actual); Study Completion 2019-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul GINESTE, PhD, Study Director — Abivax S.A.
Locations (1):
- Hospital Universitari Germans Trias i Pujol, Badalona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moron-Lopez S, Bernal S, Wong JK, Martinez-Picado J, Yukl SA. ABX464 Decreases the Total Human Immunodeficiency Virus (HIV) Reservoir and HIV Transcription Initiation in CD4+ T Cells From Antiretroviral Therapy-Suppressed Individuals Living With HIV. Clin Infect Dis. 2022 Jun 10;74(11):2044-2049. doi: 10.1093/cid/ciab733. PMID 34436569

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ABX464 150mg | ABX464 50mg for 28 Days | ABX464 50mg for 84 Days
Started | 11 | 12 | 13
Completed | 11 | 12 | 13
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ABX464 150 mg Capsules for 28 Days: ABX464 150mg: ABX464 given orally at 150 mg per day from Day 0 to Day 28 (Cohort 1/ HIV infected subjects)
- ABX464 50 mg Capsules for 28 Days: ABX464 50mg: ABX464 given orally at 50 mg per day from Day 0 to Day 28 (Cohort 2 / non HIV infected subjects)
- ABX464 50 mg Capsules for 84 Days: ABX464 50mg: ABX464 given orally at 50 mg per day from Day 0 to Day 84 (Cohort 3 / HIV infected subjects)
- Total: Total of all reporting groups
Arm/Group | ABX464 150 mg Capsules for 28 Days | ABX464 50 mg Capsules for 28 Days | ABX464 50 mg Capsules for 84 Days | Total
Number analyzed (Participants) | 11 | 12 | 13 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 12 | 13 | 36
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 11 | 12 | 13 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 11 | 12 | 13 | 36
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Spain | 11 | 12 | 13 | 36

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) of ABX464 in Sera
Description: Pharmacokinetic parameters
Time Frame: Day 1, Day 28 and Day 84
Population: Subjects who had received at least 1 dose of the Investigational Medicinal Product and who have at least baseline data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | ABX464 150mg | ABX464 50mg for 28 Days | ABX464 50mg for 84 Days
Number analyzed (Participants) | 11 | 12 | 13
ng*h/mL
  Day 1 | 306.0 (46.5) | 63.7 (39.9) | 63.7 (77.4)
  Day 28: number analyzed (Participants) | 9 | 12 | 12
  Day 28 | 119.8 (48.7) | 17.8 (60.9) | 30.3 (68.2)
  Day 84: number analyzed (Participants) | 0 | 0 | 13
  Day 84 |  |  | 28.9 (66.8)

2. Primary Outcome: Maximum Observed Concentration (Cmax) of ABX464 in Sera
Description: Pharmacokinetic parameters
Time Frame: Day 1, Day 28 and day 84
Population: Subjects who had received at least 1 dose of the Investigational Medicinal Product and who have at least baseline data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | ABX464 150mg | ABX464 50mg for 28 Days | ABX464 50mg for 84 Days
Number analyzed (Participants) | 11 | 12 | 13
ng/mL
  Day 1 | 106.1 (54.5) | 23.1 (45.2) | 24.5 (75.5)
  Day 28: number analyzed (Participants) | 9 | 12 | 13
  Day 28 | 50.9 (57.1) | 9.3 (60.3) | 13.0 (76.0)
  Day 84: number analyzed (Participants) | 0 | 0 | 12
  Day 84 |  |  | 15.6 (65.6)

3. Primary Outcome: Area Under the Curve (AUC) of ABX464 Metabolite (ABX464-N-Glucuronide) in Sera
Description: Pharmacokinetics parameters
Time Frame: Day 1, Day 28 and Day 84
Population: Subjects who had received at least 1 dose of the Investigational Medicinal Product and who have at least baseline data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- ABX461 150mg: ABX464, 50mg per Capsule Three Capsules per day for 28 days
  ABX464 150mg: ABX464 given orally at 150 mg per day from Day 0 to Day 28 (Cohort 1/ HIV infected subjects)
Arm/Group | ABX461 150mg | ABX464 50mg for 28 Days | ABX464 50mg for 84 Days
Number analyzed (Participants) | 11 | 12 | 13
ng*h/mL
  Day 1 | 50115.8 (41.5) | 8282.3 (37.0) | 11209.6 (66.5)
  Day 28: number analyzed (Participants) | 9 | 12 | 12
  Day 28 | 48605.0 (40.6) | 4800.6 (37.0) | 13308.8 (62.5)
  Day 84: number analyzed (Participants) | 0 | 0 | 12
  Day 84 |  |  | 14588.2 (58.3)

4. Primary Outcome: Maximum Observed Concentration (Cmax) of ABX464 Metabolite (ABX464-N-Glucuronide) in Sera
Description: Pharmacokinetic parameters
Time Frame: Day 1, Day 28 and Day 84
Population: Subjects who had received at least 1 dose of the Investigational Medicinal Product and who have at least baseline data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | ABX464 150mg | ABX464 50mg for 28 Days | ABX464 50mg for 84 Days
Number analyzed (Participants) | 11 | 12 | 13
ng/mL
  Day 1 | 9918.2 (33.5) | 1626.8 (36.9) | 2036.2 (62.8)
  Day 28: number analyzed (Participants) | 9 | 12 | 13
  Day 28 | 7011.1 (37.5) | 695.9 (38.6) | 1705.5 (71.8)
  Day 84: number analyzed (Participants) | 0 | 0 | 12
  Day 84 |  |  | 2150.6 (56.1)

5. Primary Outcome: Maximum Observed Concentration (Cmax) of ABX464 in Peripheral Blood Mononuclear Cells (PBMC)
Description: Pharmacokinetic parameters
Time Frame: Day 1, Day 28 and Day 84
Population: Subjects who had received at least 1 dose of the Investigational Medicinal Product and who have at least baseline data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | ABX464 150mg | ABX464 50mg for 28 Days | ABX464 50mg for 84 Days
Number analyzed (Participants) | 11 | 12 | 13
ng/mL
  Day 1 | 463.3 (55.0) | 209.4 (54.4) | 203.8 (81.0)
  Day 28: number analyzed (Participants) | 9 | 12 | 13
  Day 28 | 247.8 (75.7) | 76.4 (51.7) | 72.3 (82.9)
  Day 84: number analyzed (Participants) | 0 | 0 | 12
  Day 84 |  |  | 73.6 (57.5)

6. Primary Outcome: Area Under the Curve (AUC) of ABX464 in Peripheral Blood Mononuclear Cells (PBMC)
Description: Pharmacokinetic parameters
Time Frame: Day 1, Day 28 and Day 84
Population: Subjects who had received at least 1 dose of the Investigational Medicinal Product and who have at least baseline data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | ABX464 150mg | ABX464 50mg for 28 Days | ABX464 50mg for 84 Days
Number analyzed (Participants) | 11 | 12 | 13
ng*h/mL
  Day 1 | 1120.7 (52.6) | 594.2 (53.2) | 481.5 (78.9)
  Day 28: number analyzed (Participants) | 9 | 12 | 12
  Day 28 | 522.4 (49.2) | 156.0 (51.8) | 151.6 (74.3)
  Day 84: number analyzed (Participants) | 0 | 0 | 12
  Day 84 |  |  | 144.9 (48.6)

7. Primary Outcome: Maximum Observed Concentration (Cmax) of ABX464 Metabolite (ABX464-N-Glucuronide) in Peripheral Blood Mononuclear Cells (PBMC)
Description: Pharmacokinetic parameters
Time Frame: Day 1, Day 28 and Day 84
Population: Subjects who had received at least 1 dose of the Investigational Medicinal Product and who have at least baseline data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | ABX464 150mg | ABX464 50mg for 28 Days | ABX464 50mg for 84 Days
Number analyzed (Participants) | 11 | 12 | 13
ng/mL
  Day 1 | 585.5 (60.3) | 39.7 (90.5) | 230.0 (153.9)
  Day 28: number analyzed (Participants) | 9 | 12 | 13
  Day 28 | 491.5 (73.0) | 35.6 (85.7) | 125.1 (86.1)
  Day 84: number analyzed (Participants) | 0 | 0 | 12
  Day 84 |  |  | 153.3 (49.4)

8. Primary Outcome: Area Under the Curve (AUC) of ABX464 Metabolite (ABX464-N-Glucuronide) in Peripheral Blood Mononuclear Cells (PBMC)
Description: Pharmacokinetic parameters
Time Frame: Day 1, Day 28 and Day 84
Population: Subjects who had received at least 1 dose of the Investigational Medicinal Product and who have at least baseline data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | ABX464 150mg | ABX464 50mg for 28 Days | ABX464 50mg for 84 Days
Number analyzed (Participants) | 11 | 12 | 13
ng*h/mL
  Day 1 | 2133.7 (42.2) | 39.2 (186.7) | 835.3 (116.0)
  Day 28: number analyzed (Participants) | 9 | 12 | 12
  Day 28 | 2212.3 (58.8) | 35.0 (210.1) | 697.5 (92.0)
  Day 84: number analyzed (Participants) | 0 | 0 | 12
  Day 84 |  |  | 766.5 (57.4)

9. Primary Outcome: Concentration of ABX464 in Rectal Tissue (Measured Only at Pre-infusion Timepoint)
Description: Pharmacokinetic parameters
Time Frame: Day 1, Day 28, Day 56, Day 84 and Day 112
Population: Subjects who had received at least 1 dose of the Investigational Medicinal Product and who have at least baseline data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ABX464 150mg | ABX464 50mg for 28 Days | ABX464 50mg for 84 Days
Number analyzed (Participants) | 11 | 12 | 13
ng/mL
  Day 1: number analyzed (Participants) | 11 | 12 | 12
  Day 1 | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Day 28: number analyzed (Participants) | 8 | 12 | 11
  Day 28 | 0.1 (0.11) | 0.1 (0.19) | 0.1 (0.13)
  Day 56: number analyzed (Participants) | 10 | 0 | 0
  Day 56 | 0.0 (0.00) |  |
  Day 84: number analyzed (Participants) | 0 | 0 | 12
  Day 84 |  |  | 0.1 (0.13)
  Day 112: number analyzed (Participants) | 0 | 0 | 12
  Day 112 |  |  | 0.0 (0.00)

10. Primary Outcome: Concentration of ABX464 Metabolite (ABX464-N-Glucuronide) in Rectal Tissue (Measured Only at Pre-infusion Timepoint)
Description: Pharmacokinetic parameters
Time Frame: Day 1, Day 28, Day 56, Day 84 and Day 112
Population: Subjects who had received at least 1 dose of the Investigational Medicinal Product and who have at least baseline data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ABX464 150mg | ABX464 50mg for 28 Days | ABX464 50mg for 84 Days
Number analyzed (Participants) | 11 | 12 | 12
ng/mL
  Day 1 | 0.0 (0.00) | 0.1 (0.08) | 0.0 (0.00)
  Day 28: number analyzed (Participants) | 8 | 12 | 11
  Day 28 | 0.1 (0.04) | 0.1 (0.11) | 0.1 (0.09)
  Day 56: number analyzed (Participants) | 10 | 0 | 0
  Day 56 | 0.0 (0.00) |  |
  Day 84: number analyzed (Participants) | 0 | 0 | 12
  Day 84 |  |  | 0.2 (0.11)
  Day 112: number analyzed (Participants) | 0 | 0 | 12
  Day 112 |  |  | 0.0 (0.00)

11. Secondary Outcome: Mean Change From Baseline in Plasma Viral Load (Ultrasensitive Assay)
Description: Viral Load Assessments (HIV-1 RNA copies/ml)
Time Frame: Day 28, Day 56, Day 84 and Day 112
Population: Subjects who had received at least 1 dose of the Investigational Medicinal Product and who have at least baseline data. HIV viral measurements were not assessed for cohort 2 subjects as they were HIV non infected subjets.
Measure: Mean (95% Confidence Interval); unit: copies/mL
Groups:
- ABX464 50mg: ABX464, 50mg per Capsule One Capsule per day for 84 days
  ABX464 50mg: ABX464 given orally at 50 mg per day from Day 0 to Day 84 (Cohort 3 / HIV infected subjects)
Arm/Group | ABX464 150mg | ABX464 50mg
Number analyzed (Participants) | 9 | 8
copies/mL
  Day 28 | -0.9 [-1.9 to 0.1] | -2.0 [-4.3 to 0.2]
  Day 56: number analyzed (Participants) | 9 | 0
  Day 56 | -0.4 [-1.5 to 0.7] |
  Day 84: number analyzed (Participants) | 0 | 8
  Day 84 |  | -0.9 [-3.0 to 1.2]
  Day 112: number analyzed (Participants) | 0 | 8
  Day 112 |  | -1.1 [-3.7 to 1.5]

12. Secondary Outcome: CD4+ Counts (Cell/mm^3)
Description: T-cell determinations
Time Frame: Day 28, Day 35, Day 56, Day 84, Day 91 and Day 112
Population: Subjects who had received at least 1 dose of the Investigational Medicinal Product and who have at least baseline data. CD4+ counts measurements were not assessed for cohort 2 subjects as they were HIV non infected subjets.
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | ABX464 150mg | ABX464 50mg
Number analyzed (Participants) | 9 | 12
cells/mm^3
  Day 28 | -130.6 [-217.5 to -43.6] | -34.6 [-167.7 to 98.5]
  Day 35: number analyzed (Participants) | 9 | 0
  Day 35 | -125.6 [-266.2 to 15.1] |
  Day 56: number analyzed (Participants) | 9 | 0
  Day 56 | 29.6 [-202.4 to 261.5] |
  Day 84: number analyzed (Participants) | 0 | 12
  Day 84 |  | 8.3 [-90.2 to 106.9]
  Day 91: number analyzed (Participants) | 0 | 12
  Day 91 |  | 23.3 [-122.5 to 169.0]
  Day 112: number analyzed (Participants) | 0 | 12
  Day 112 |  | 161.8 [59.5 to 264.2]

13. Secondary Outcome: Total HIV-1 DNA Reservoir in Peripheral Blood Mononuclear Cells (PBMC)
Description: HIV reservoir cells (CD4+)
Time Frame: Day 28, Day 56, Day 84 and Day 112
Population: Subjects who had received at least 1 dose of the Investigational Medicinal Product and who have at least baseline data. Total HIV-1 DNA reservoir measurements were not assessed for cohort 2 subjects as they were HIV non infected subjets.
Measure: Mean (95% Confidence Interval); unit: copies/10^6 cells
Arm/Group | ABX464 150mg | ABX464 50mg
Number analyzed (Participants) | 9 | 12
copies/10^6 cells
  Day 28 | -86.8 [-172.2 to -1.3] | 22.3 [-21.7 to 66.4]
  Day 56: number analyzed (Participants) | 9 | 0
  Day 56 | -37.1 [-139.1 to 64.9] |
  Day 84: number analyzed (Participants) | 0 | 12
  Day 84 |  | 10.8 [-55.3 to 76.9]
  Day 112: number analyzed (Participants) | 0 | 12
  Day 112 |  | 95.6 [26.1 to 165.0]

ADVERSE EVENTS:
Time Frame: From baseline up to 112 days
Description: Subjects who had received at least 1 dose of the Investigational Medicinal Product and who have at least baseline data.
Arm/Group | ABX464 150mg | ABX464 50mg for 28 Days | ABX464 50mg for 84 Days
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 9/11 | 3/12 | 7/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABX464 150mg (N=11) | ABX464 50mg for 28 Days (N=12) | ABX464 50mg for 84 Days (N=13)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 0 (0) | 2 (2)
Asthemia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperamylasaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperlipaseamia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 8 (9) | 2 (2) | 4 (4)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (5) | 0 (0) | 1 (2)
Thirst (General disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Nightmare (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-09-04): https://cdn.clinicaltrials.gov/large-docs/25/NCT02990325/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-29): https://cdn.clinicaltrials.gov/large-docs/25/NCT02990325/SAP_001.pdf